CLINICAL TRIAL: NCT04220528
Title: Single Arm, Open, Multicenter Phase II Clinical Study of Radical Radiotherapy and Chemotherapy Combined With Maintenance Chemotherapy in the Treatment of Stage N3 NPC
Brief Title: Radical Radiotherapy and Chemotherapy Combined With Maintenance Chemotherapy in the Treatment of Stage N3 NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Jiangxi Provincial Cancer Hospital (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC002.1
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radical chemoradiotherapy plus oral capecitabine/teggiol (Experimental): Patients with newly diagnosed, non-metastatic stage N3 NPC was given Teggio 40-60mg bid d1-14, q4w, oral maintenance chemotherapy for 1 year or capecitabine 2500mg/m2/d twice daily oral d1-14, q4w after receiving radical chemoradiotherapy.
  Interventions: Drug: Capecitabine/Tiggio

INTERVENTIONS:
Drug: Capecitabine/Tiggio — Drug: Capecitabine/Tiggio
  Radical chemoradiotherapy：Induction chemotherapy plus Concurrent chemoradiotherapy
  Induction chemotherapy：Gemcitabine (1000mg/m2) D1 D8+ nida platinum (80mg/m2) D2 q3w ×3cycle
  Concurrent chemoradiotherapy：IMRT was used for radiotherapy, during which D1 and D22 were given two cycles of single drug concurrent chemotherapy with nidapatin (100mg/m2).
  Other Names: Radiation

SUMMARY:
This study is a randomized, phase II, prospective, multicenter clinical trial to evaluate the efficacy and safety of radical chemoradiotherapy plus oral capecitabine/teggio for 1 year in patients with N3.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis (pathologically confirmed by nasopharyngeal biopsy) was nasopharyngeal carcinoma;
2. No distant metastatic stage N3 nasopharyngeal carcinoma was first diagnosed (according to the 8th edition UICC/AJCC nasopharyngeal carcinoma staging system defined as any T and N3M0 stage nasopharyngeal carcinoma).
3. Aged 18-65;
4. At least one measurable tumor lesion;
5. PS (ECOG standard) 0-1;
6. Adequate hematopoietic function: WBC≥3.5×109/L, Hb≥100g/L, PLT≥100×109/L;
7. Normal liver and kidney functions: ALT/AST < 2.5 times the upper limit of normal value (ULN), total bilirubin < 1.5×ULN;Serum creatinine < 1.5×ULN;
8. Expected survival period ≥6 months;
9. Signing informed consent;
10. Follow up regularly and comply with test requirements.

Exclusion Criteria:

1. Patients with distant organ metastasis;
2. Recurrent nasopharyngeal carcinoma;
3. Creatinine clearance rate <60ml/ min;
4. Have received chemotherapy, radiotherapy or targeted therapy;
5. Have or are suffering from other malignant tumors within 5 years (except non-melanoma skin cancer or pre-invasive cervical cancer);
6. Serious complications, such as uncontrolled hypertension, coronary heart disease, diabetes, heart failure, etc.
7. Active systemic infection;
8. History of serious lung or heart disease;
9. Drug or alcohol abuse;
10. No or limited capacity for civil conduct;
11. The patient has a physical or mental disorder, and the researcher considers that the patient is unable to fully or fully understand the possible complications of this study;
12. Receive chronic systemic immunotherapy or hormone therapy outside the study;
13. Pregnancy or lactation period;
14. Patients receive blind treatment in other clinical studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) | 24 months
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China